CLINICAL TRIAL: NCT06420817
Title: Effect of a Customised Lifestyle Medicine Strategy on Lowering Blood Lipid Levels in Indian Physicians
Acronym: CLIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Collaborators: Christian Medical College, Vellore, India (Other)
Responsible Party: Principal Investigator, Dr. Manoj Varanattu, Professor of Pediatrics & Neonatology, Jubilee Mission Medical College and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CLIP
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Lifestyle Risk Reduction; Cholesterol, Elevated; LDL Hyperlipoproteinemia; Hypertension; Lipoprotein(A); HbA1C; BMI
Keywords: Intermittend fasting; Blood lipid level lowering
MeSH Terms: conditions — Risk Reduction Behavior; Hypercholesterolemia; Hypertension | interventions — Exercise; Post-Exercise Recovery

STUDY DESIGN:
Intervention Model Description: The study would be done in 2 phases. In the first phase the pretest questionnaire would be administered throughGoogle forms and health education on various Lifestyle Medicine interventions would be given. In the second phase Intervention would be carried out and monitoring would be done online daily / weekly by the investigative team.
  The following five strategies of lifestyle medicine will be tried to lower the lipid levels in the study group:
  1. Nutrition - modified/Indianized Portfolio diet - (Primary Intervention)
  2. adequate exercise - 180 minutes of moderate intensity exercises every week
  3. intermittent fasting of 12 hours every day
  4. sleep monitoring and
  5. monitoring stress levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Interventions (Experimental): Lifestyle Interventions (a prescribed whole food plant-based diet, physical activity and intermittent fasting along with monitoring of sleep and stress levels) would be carried out to the enrolled participants
  Interventions: Behavioral: Indian version of a 'Portfolio' diet; Behavioral: Physical Activity; Behavioral: Intermittent fasting; Behavioral: Monitoring of sleep and stress levels

INTERVENTIONS:
Behavioral: Indian version of a 'Portfolio' diet — The participants will be required to follow the prescribed diet plan for 4 weeks
  Other Names: Indian version of a dietary portfolio of cholesterol lowering foods
Behavioral: Physical Activity — The participants will be required to join for an hour of group online exercise program 3 days a week for 4 weeks
  • (Exercise Duration = 180 minutes per week including cardio, strength training and flexibility)
  Other Names: Exercise; Workout
Behavioral: Intermittent fasting — The participants will be required to do intermittent fasting for 12 hours daily for 4 weeks
  Other Names: Time Restricted Eating
Behavioral: Monitoring of sleep and stress levels — The participants will be required to monitor their sleep and stress levels

SUMMARY:
Lifestyle medicine is a medical specialty that uses evidence-based therapeutic interventions to prevent, treat, and reverse chronic conditions. Studies have shown that a 50 mg/dl reduction in LDL reduces the risk of developing stroke by 20%, and a 10 mm Hg reduction in systolic BP reduces the risk of developing MACE by 22% and stroke by 41%. The CLIP (Cholesterol Lowering Lifestyle Intervention Project) is an innovative initiative proposed to evaluate the combined effect of an Indian version of Portfolio diet-based nutrition strategy, intermittent fasting, exercise, sleep, and stress reduction techniques on lowering blood lipid levels in health professionals and their family. The study aims to evaluate the effect of CLIP on changes in blood pressure, weight, HbA1C levels, blood CRP levels, and other blood parameters.

DETAILED DESCRIPTION:
Lifestyle medicine is a medical specialty that uses evidence based therapeutic lifestyle interventions as a primary modality to prevent, treat and often reverse chronic conditions using whole food plant-based diet, physical activity, restorative sleep, stress reduction, avoiding risky substances and positive social connections with or without medications.

Epidemiological and interventional studies have shown clearly that a 50 mg/dl reduction in LDL reduces the risk of developing stroke by 20% and a 10 mm Hg reduction in systolic BP reduces the risk of developing MACE by 22% and the risk of developing stroke by 41%.(Enas EA, et al, Indian Heart Journal, 2011, cadiresearch.org,) Studies by the nutrition expert David J.A. Jenkins and colleagues from Toronto University have shown that grouping plant based whole foods, which have their own cholesterol lowering ability when eaten alone, will have a larger effect when they are eaten together or combined into a "portfolio" as part of a regular diet (https://jamanetwork.com/journals/jama/fullarticle /196970). The 'portfolio diet' plan has been subsequently shown to reduce cholesterol similar to powerful cholesterol-lowering drugs without any side effects in various other studies as well. However, no study has so far looked at the effects of this diet on Indian population. Also, no reported study in the world so far has looked at the effects of a combination of lifestyle medicine interventions including the Indianized version of portfolio diet on the reduction of lipid levels in health care workers CLIP (Cholesterol lowering Lifestyle Intervention Project) is an innovative lifestyle medicine intervention project that we propose to carry out under the academic guidance of the Dept of Lifestyle Medicine , CMC, Vellore.

Research Question: Will a customised lifestyle medicine strategy over a period of 4 weeks lower blood lipid levels significantly in adults between 18 and 70 years?

Null Hypothesis: A customised lifestyle medicine strategy over a period of 4 weeks will not significantly lower blood lipid levels in adults between 18 and 70 years Type of study: A Quasi Experimental Study

Time duration:

Preparation: 4 weeks Intervention: 4 weeks Result compilation and analysis: 4 months Total: 6 months

AIM: To evaluate the combined effect of an Indian version of Portfolio diet-based nutrition strategy, Intermittent fasting, Exercise, Sleep and Stress Reduction Techniques on lowering blood lipid levels in health professionals and their family

Secondary objectives: To evaluate the effect of the CLIP interventions on the changes in

* Blood Pressure
* Weight
* HbA1C levels
* Blood CRP levels
* Other blood Parameters including Lipo A

The study would be done in 2 phases. In the first phase the pretest questionnaire would be administered through google forms and health education on whole food plant-based diet, physical activity, restorative sleep, stress reduction & avoiding risky substances would be given.

In the second phase Intervention would be carried out and monitoring would be done online daily / weekly by the investigative team.

Population: Willing members of health professionals and their family Inclusion Criteria: All willing health professionals and their family aged between 18 and 70 years

Exclusion Criteria:

* Those who have been started on any medication for chronic illnesses unless sufficient period (3 months) is over for stabilization of parameters on those medications.
* People on insulin, steroids and warfarin.
* Those who alter their medications during the intervention
* Those who are unfit to exercise

Methods:

Enrolment and Training:

All the participants who meet the criteria for the study will be enrolled from an already existing WhatsApp group of Modern Medicine doctors and their family interested in lifestyle interventions.

The study protocol will be familiarised online through social media platforms on the basic concepts of lifestyle medicine in general and the interventions adopted in particular, before the commencement of the intervention.

Consenting members will be enrolled in the study and will undergo the following interventions:

I. Baseline Screening: The following parameters will be evaluated (by the participants) during the preparation stage before the commencement of the intervention:

Anthropometry & Clinical: Height, Weight, Waist Circumference, Waist to Hip Ratio, BP Biochemistry: Lipid Profile, Apolipoprotein B, Lipoprotein A, HbA1C, Blood sugar (Fasting and PP), CRP, LFT, RFT, Uric Acid, TSH

II. Lifestyle Interventions: The participants will be supervised to

* follow the prescribed diet plan
* do intermittent fasting for 12 hours daily and
* join for an hour of group online exercise program 3 days a week.
* Monitor the sleep duration as per PSQI (Pittsburgh sleep quality index) scores
* (Exercise Duration = 180 minutes per week including cardio, strength training and flexibility)
* Compliance: Adherence to all interventions planned will be monitored through a weekly questionnaire, software like habit tracker and online Zoom meetings

III. Final Evaluation: Final Anthropometry, Clinical and Biochemical Parameters achieved will be obtained at the end of 4 weeks. (Pre and post biochemical evaluation will be done by the participants in the same lab)

Expected outcome of the study: It is expected that diet and other lifestyle interventions included in the study will lower total cholesterol and LDL levels (primary outcomes) of the participants in proportion to their degree of compliance to interventions.

1. Proportion of participants achieving reduction in BMI & Waist to Hip Ratio
2. Proportion of hypertensive participants achieving reduction in BP
3. Proportion of DM participants achieving reduction in HbA1C
4. Proportion of participants achieving reduction in TC & LDL levels
5. Proportion of participants achieving reduction in all the other biochemical parameters studied

ELIGIBILITY:
Inclusion Criteria: All willing Indian doctors and their family aged between 18 and 70 years

Exclusion Criteria:

* Those who have been started on any medication for chronic illnesses unless sufficient period (3 months) is over for stabilization of parameters on those medications.
* People on insulin, steroids and warfarin.
* Those who alter their medications during the intervention
* Those who are unfit to exercise

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Changes in the blood lipid levels | 4 weeks
  The combined effect of an Indian version of Portfolio diet-based nutrition strategy, Intermittent fasting, Exercise, Sleep and Stress Reduction Techniques on lowering blood lipid levels

SECONDARY OUTCOMES:
Changes in the anthropometric and biochemical parameters | 4 weeks
  The effect of a customised lifestyle intervention technique on changes in Blood Pressure, Weight, BMI, HbA1C levels, Blood HS CRP levels and Other blood Parameters including Lipoprotein A

CONTACTS AND LOCATIONS:
Locations (1):
- Manoj Varanattu, Thrissur, Kerala, India

REFERENCES:
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Wong JM, de Souza R, Emam A, Parker TL, Vidgen E, Trautwein EA, Lapsley KG, Josse RG, Leiter LA, Singer W, Connelly PW. Direct comparison of a dietary portfolio of cholesterol-lowering foods with a statin in hypercholesterolemic participants. Am J Clin Nutr. 2005 Feb;81(2):380-7. doi: 10.1093/ajcn.81.2.380. PMID 15699225
- [Background] Khodamoradi K, Khosropanah MH, Ayati Z, Chang D, Nasli-Esfahani E, Ayati MH, Namazi N. The Effects of Fenugreek on Cardiometabolic Risk Factors in Adults: A Systematic Review and Meta-analysis. Complement Ther Med. 2020 Aug;52:102416. doi: 10.1016/j.ctim.2020.102416. Epub 2020 Apr 28. PMID 32951700
- [Background] Heshmat-Ghahdarijani K, Mashayekhiasl N, Amerizadeh A, Teimouri Jervekani Z, Sadeghi M. Effect of fenugreek consumption on serum lipid profile: A systematic review and meta-analysis. Phytother Res. 2020 Sep;34(9):2230-2245. doi: 10.1002/ptr.6690. Epub 2020 May 8. PMID 32385866
- [Background] Gopa B, Bhatt J, Hemavathi KG. A comparative clinical study of hypolipidemic efficacy of Amla (Emblica officinalis) with 3-hydroxy-3-methylglutaryl-coenzyme-A reductase inhibitor simvastatin. Indian J Pharmacol. 2012 Mar;44(2):238-42. doi: 10.4103/0253-7613.93857. PMID 22529483
- [Background] Akhtar MS, Ramzan A, Ali A, Ahmad M. Effect of Amla fruit (Emblica officinalis Gaertn.) on blood glucose and lipid profile of normal subjects and type 2 diabetic patients. Int J Food Sci Nutr. 2011 Sep;62(6):609-16. doi: 10.3109/09637486.2011.560565. Epub 2011 Apr 18. PMID 21495900
- [Background] Uma Maheswari K, Dilara K, Vadivel S, Johnson P, Jayaraman S. A review on hypo-cholesterolemic activity of Nigella sativa seeds and its extracts. Bioinformation. 2022 Apr 30;18(4):343-348. doi: 10.6026/97320630018343. eCollection 2022. PMID 36909699
- [Background] Hallajzadeh J, Milajerdi A, Mobini M, Amirani E, Azizi S, Nikkhah E, Bahadori B, Sheikhsoleimani R, Mirhashemi SM. Effects of Nigella sativa on glycemic control, lipid profiles, and biomarkers of inflammatory and oxidative stress: A systematic review and meta-analysis of randomized controlled clinical trials. Phytother Res. 2020 Oct;34(10):2586-2608. doi: 10.1002/ptr.6708. Epub 2020 May 11. PMID 32394508
- [Background] Sahebkar A, Beccuti G, Simental-Mendia LE, Nobili V, Bo S. Nigella sativa (black seed) effects on plasma lipid concentrations in humans: A systematic review and meta-analysis of randomized placebo-controlled trials. Pharmacol Res. 2016 Apr;106:37-50. doi: 10.1016/j.phrs.2016.02.008. Epub 2016 Feb 10. PMID 26875640
- [Background] Prasad K, Khan AS, Shoker M. Flaxseed and Its Components in Treatment of Hyperlipidemia and Cardiovascular Disease. Int J Angiol. 2020 Dec;29(4):216-222. doi: 10.1055/s-0040-1709129. Epub 2020 Apr 14. PMID 33268971
- [Background] Sadat Masjedi M, Mohammadi Pour P, Shokoohinia Y, Asgary S. Effects of Flaxseed on Blood Lipids in Healthy and Dyslipidemic Subjects: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Curr Probl Cardiol. 2022 Jul;47(7):100931. doi: 10.1016/j.cpcardiol.2021.100931. Epub 2021 Jul 16. PMID 34384619
- [Background] Amiri M, Raeisi-Dehkordi H, Sarrafzadegan N, Forbes SC, Salehi-Abargouei A. The effects of Canola oil on cardiovascular risk factors: A systematic review and meta-analysis with dose-response analysis of controlled clinical trials. Nutr Metab Cardiovasc Dis. 2020 Nov 27;30(12):2133-2145. doi: 10.1016/j.numecd.2020.06.007. Epub 2020 Jun 18. PMID 33127255
- [Background] Schwingshackl L, Bogensberger B, Bencic A, Knuppel S, Boeing H, Hoffmann G. Effects of oils and solid fats on blood lipids: a systematic review and network meta-analysis. J Lipid Res. 2018 Sep;59(9):1771-1782. doi: 10.1194/jlr.P085522. Epub 2018 Jul 13. PMID 30006369
- [Background] Wilson TA, Ausman LM, Lawton CW, Hegsted DM, Nicolosi RJ. Comparative cholesterol lowering properties of vegetable oils: beyond fatty acids. J Am Coll Nutr. 2000 Oct;19(5):601-7. doi: 10.1080/07315724.2000.10718957. PMID 11022873
- [Background] Saedi S, Noroozi M, Khosrotabar N, Mazandarani S, Ghadrdoost B. How canola and sunflower oils affect lipid profile and anthropometric parameters of participants with dyslipidemia. Med J Islam Repub Iran. 2017 Jan 15;31:5. doi: 10.18869/mjiri.31.5. eCollection 2017. PMID 28638812
- [Background] Craig WJ, Mangels AR, Fresan U, Marsh K, Miles FL, Saunders AV, Haddad EH, Heskey CE, Johnston P, Larson-Meyer E, Orlich M. The Safe and Effective Use of Plant-Based Diets with Guidelines for Health Professionals. Nutrients. 2021 Nov 19;13(11):4144. doi: 10.3390/nu13114144. PMID 34836399
- [Background] Sabate J, Oda K, Ros E. Nut consumption and blood lipid levels: a pooled analysis of 25 intervention trials. Arch Intern Med. 2010 May 10;170(9):821-7. doi: 10.1001/archinternmed.2010.79. PMID 20458092
- [Background] Liu AG, Ford NA, Hu FB, Zelman KM, Mozaffarian D, Kris-Etherton PM. A healthy approach to dietary fats: understanding the science and taking action to reduce consumer confusion. Nutr J. 2017 Aug 30;16(1):53. doi: 10.1186/s12937-017-0271-4. PMID 28854932
- [Background] Zhang Z, Lanza E, Kris-Etherton PM, Colburn NH, Bagshaw D, Rovine MJ, Ulbrecht JS, Bobe G, Chapkin RS, Hartman TJ. A high legume low glycemic index diet improves serum lipid profiles in men. Lipids. 2010 Sep;45(9):765-75. doi: 10.1007/s11745-010-3463-7. Epub 2010 Aug 24. PMID 20734238
- [Background] Ha V, Sievenpiper JL, de Souza RJ, Jayalath VH, Mirrahimi A, Agarwal A, Chiavaroli L, Mejia SB, Sacks FM, Di Buono M, Bernstein AM, Leiter LA, Kris-Etherton PM, Vuksan V, Bazinet RP, Josse RG, Beyene J, Kendall CW, Jenkins DJ. Effect of dietary pulse intake on established therapeutic lipid targets for cardiovascular risk reduction: a systematic review and meta-analysis of randomized controlled trials. CMAJ. 2014 May 13;186(8):E252-62. doi: 10.1503/cmaj.131727. Epub 2014 Apr 7. PMID 24710915
- [Background] Schoeneck M, Iggman D. The effects of foods on LDL cholesterol levels: A systematic review of the accumulated evidence from systematic reviews and meta-analyses of randomized controlled trials. Nutr Metab Cardiovasc Dis. 2021 May 6;31(5):1325-1338. doi: 10.1016/j.numecd.2020.12.032. Epub 2021 Jan 16. PMID 33762150
- [Background] Richter CK, Skulas-Ray AC, Champagne CM, Kris-Etherton PM. Plant protein and animal proteins: do they differentially affect cardiovascular disease risk? Adv Nutr. 2015 Nov 13;6(6):712-28. doi: 10.3945/an.115.009654. Print 2015 Nov. PMID 26567196
- [Background] Erdman JW Jr. AHA Science Advisory: Soy protein and cardiovascular disease: A statement for healthcare professionals from the Nutrition Committee of the AHA. Circulation. 2000 Nov 14;102(20):2555-9. doi: 10.1161/01.cir.102.20.2555. No abstract available. PMID 11076833
- [Background] Yu-Poth S, Zhao G, Etherton T, Naglak M, Jonnalagadda S, Kris-Etherton PM. Effects of the National Cholesterol Education Program's Step I and Step II dietary intervention programs on cardiovascular disease risk factors: a meta-analysis. Am J Clin Nutr. 1999 Apr;69(4):632-46. doi: 10.1093/ajcn/69.4.632. PMID 10197564
- [Background] Anderson JW, Johnstone BM, Cook-Newell ME. Meta-analysis of the effects of soy protein intake on serum lipids. N Engl J Med. 1995 Aug 3;333(5):276-82. doi: 10.1056/NEJM199508033330502. PMID 7596371
- [Background] Teixeira SR, Potter SM, Weigel R, Hannum S, Erdman JW Jr, Hasler CM. Effects of feeding 4 levels of soy protein for 3 and 6 wk on blood lipids and apolipoproteins in moderately hypercholesterolemic men. Am J Clin Nutr. 2000 May;71(5):1077-84. doi: 10.1093/ajcn/71.5.1077. PMID 10799368
- [Background] Chiavaroli L, Nishi SK, Khan TA, Braunstein CR, Glenn AJ, Mejia SB, Rahelic D, Kahleova H, Salas-Salvado J, Jenkins DJA, Kendall CWC, Sievenpiper JL. Portfolio Dietary Pattern and Cardiovascular Disease: A Systematic Review and Meta-analysis of Controlled Trials. Prog Cardiovasc Dis. 2018 May-Jun;61(1):43-53. doi: 10.1016/j.pcad.2018.05.004. Epub 2018 May 26. PMID 29807048
- [Background] Li SS, Blanco Mejia S, Lytvyn L, Stewart SE, Viguiliouk E, Ha V, de Souza RJ, Leiter LA, Kendall CWC, Jenkins DJA, Sievenpiper JL. Effect of Plant Protein on Blood Lipids: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2017 Dec 20;6(12):e006659. doi: 10.1161/JAHA.117.006659. PMID 29263032
- [Background] Reddy KR, Freeman AM. Lifestyle Medicine: An Antidote to Cardiovascular Diseases. Am J Lifestyle Med. 2022 Oct 3;18(2):216-232. doi: 10.1177/15598276221130684. eCollection 2024 Mar-Apr. PMID 38559785
- [Background] Lo K, Glenn AJ, Yeung S, Kendall CWC, Sievenpiper JL, Jenkins DJA, Woo J. Prospective Association of the Portfolio Diet with All-Cause and Cause-Specific Mortality Risk in the Mr. OS and Ms. OS Study. Nutrients. 2021 Dec 3;13(12):4360. doi: 10.3390/nu13124360. PMID 34959911
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Wong JM, de Souza R, Emam A, Parker TL, Vidgen E, Lapsley KG, Trautwein EA, Josse RG, Leiter LA, Connelly PW. Effects of a dietary portfolio of cholesterol-lowering foods vs lovastatin on serum lipids and C-reactive protein. JAMA. 2003 Jul 23;290(4):502-10. doi: 10.1001/jama.290.4.502. PMID 12876093
- [Background] Wang Y, Xu D. Effects of aerobic exercise on lipids and lipoproteins. Lipids Health Dis. 2017 Jul 5;16(1):132. doi: 10.1186/s12944-017-0515-5. PMID 28679436
- [Background] Muscella A, Stefano E, Marsigliante S. The effects of exercise training on lipid metabolism and coronary heart disease. Am J Physiol Heart Circ Physiol. 2020 Jul 1;319(1):H76-H88. doi: 10.1152/ajpheart.00708.2019. Epub 2020 May 22. PMID 32442027
- [Background] Smiley A, King D, Harezlak J, Dinh P, Bidulescu A. The association between sleep duration and lipid profiles: the NHANES 2013-2014. J Diabetes Metab Disord. 2019 Jun 22;18(2):315-322. doi: 10.1007/s40200-019-00415-0. eCollection 2019 Dec. PMID 31890656
- [Background] Makarem N, Castro-Diehl C, St-Onge MP, Redline S, Shea S, Lloyd-Jones D, Ning H, Aggarwal B. Redefining Cardiovascular Health to Include Sleep: Prospective Associations With Cardiovascular Disease in the MESA Sleep Study. J Am Heart Assoc. 2022 Nov;11(21):e025252. doi: 10.1161/JAHA.122.025252. Epub 2022 Oct 19. PMID 36259552
- [Background] Zhang J, Zhang J, Wu H, Wang R. Sleep duration and risk of hyperlipidemia: a systematic review and meta-analysis of prospective studies. Sleep Breath. 2022 Sep;26(3):997-1010. doi: 10.1007/s11325-021-02504-y. Epub 2021 Oct 7. PMID 34618292
- [Background] Assadi SN. What are the effects of psychological stress and physical work on blood lipid profiles? Medicine (Baltimore). 2017 May;96(18):e6816. doi: 10.1097/MD.0000000000006816. PMID 28471984
- [Background] Kivimaki M, Steptoe A. Effects of stress on the development and progression of cardiovascular disease. Nat Rev Cardiol. 2018 Apr;15(4):215-229. doi: 10.1038/nrcardio.2017.189. Epub 2017 Dec 7. PMID 29213140
- [Background] Sara JD, Prasad M, Eleid MF, Zhang M, Widmer RJ, Lerman A. Association Between Work-Related Stress and Coronary Heart Disease: A Review of Prospective Studies Through the Job Strain, Effort-Reward Balance, and Organizational Justice Models. J Am Heart Assoc. 2018 Apr 27;7(9):e008073. doi: 10.1161/JAHA.117.008073. No abstract available. PMID 29703810